CLINICAL TRIAL: NCT02811419
Title: I-scan Versus Standard High-Definition White Light for the Detection of Adenomatous Polyps
Brief Title: I-scan for Adenoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P072016
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Adenomatous Polyps
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- i-scan (Active Comparator): Inspection with i-scan surface enhancement
  Interventions: Device: i-scan
- Standard high-definition white light (Active Comparator): Inspection with standard high-definition white light (usual care)
  Interventions: Device: standard high-definition white light

INTERVENTIONS:
Device: i-scan — examination will be performed with i-scan digital enhancement
  Other Names: colonoscopy
  Arms: i-scan
Device: standard high-definition white light — examination will be performed with high-definition white light
  Other Names: colonoscopy
  Arms: Standard high-definition white light

SUMMARY:
This study is a randomized controlled trial to determine whether i-scan can improve the detection of conventional adenomas and sessile serrated adenomas/polyps.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing the use of i-scan (digital surface and contrast enhancement of the mucosa) versus standard high-definition white light for the detection of conventional adenomas and sessile serrated adenomas/polyps. Recent studies have indicated that colonoscopy is more effective in preventing cancer in the left side of the colon than the right side of the colon. The reasons for this difference may be partly biologic, in that a special group of polyps known as sessile serrated adenomas/polyps (SSA) are located primarily proximal to the splenic flexure. Sessile serrated adenomas/polyps share molecular features with a group of cancers that occur primarily in the proximal colon. These molecular features include CpG island methylator phenotype (CIMP) and microsatellite instability. These lesions are endoscopically subtle in that they are often flat, have the same color as the surrounding mucosa, and are hard to differentiate from normal mucosa. Recent studies have shown that image enhanced endoscopy can highlight the appearance of these lesions. This study will test whether i-scan increases the detection of conventional adenomas and sessile serrated adenomas/polyps in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75
* Intact colon and rectum
* Willing to sign an informed consent form

Exclusion Criteria:

* Subjects less than 50 years of age or greater than 75 years of age
* Subjects who are in the inpatient unit
* Subjects with diverticulitis,
* Subjects with inflammatory bowel disease
* Subjects with polyposis syndromes
* Subjects with previous surgical resection of any portion of the colon or rectum
* Subjects referred for endoscopic resection of previously diagnosed colorectal polyp

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey K Lee, MD, Principal Investigator — Primary
Locations (1):
- University of California San Francisco Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kidambi TD, Terdiman JP, El-Nachef N, Singh A, Kattah MG, Lee JK. Effect of I-scan Electronic Chromoendoscopy on Detection of Adenomas During Colonoscopy. Clin Gastroenterol Hepatol. 2019 Mar;17(4):701-708.e1. doi: 10.1016/j.cgh.2018.06.024. Epub 2018 Jun 20. PMID 29935326

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention (I-scan): i-scan 1 (surface enhancement with contrast enhancement)
- Control (HDWL): HDWL (High definition white light)
Period: Overall Study
Arm/Group | Intervention (I-scan) | Control (HDWL)
Started | 369 | 371
Completed | 357 | 358
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I-scan | Standard High-definition White Light | Total
Number analyzed (Participants) | 369 | 371 | 740
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (7.5) | 60.8 (7.5) | 61.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 187 | 372
  Male | 184 | 184 | 368
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 369 | 371 | 740
Region of Enrollment [Number; unit: participants]
  United States | 369 | 371 | 740
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (5.7) | 26.5 (4.9) | 26.7 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Conventional Adenoma and Sessile Serrated Adenoma/Polyp Detected
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (I-scan) | Control (HDWL)
Number analyzed (Participants) | 369 | 371
Participants | 208 | 171

2. Secondary Outcome: Number of Participants With Conventional Adenoma Detected
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (I-scan) | Control (HDWL)
Number analyzed (Participants) | 369 | 371
Participants | 174 | 140

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention (I-scan) | Control (HDWL)
All-Cause Mortality (participants affected / at risk) | 0/369 | 0/371
Serious Adverse Events (participants affected / at risk) | 0/369 | 0/371
Other Adverse Events (participants affected / at risk) | 0/369 | 0/371

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT02811419/Prot_SAP_000.pdf